CLINICAL TRIAL: NCT03122678
Title: Thiamine Supplementation in Patients With Septic Shock: A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Thiamine Supplementation in Patients With Septic Shock
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participant enrolled
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Jinesh Mehta, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLA 16-058
Record Dates: First submitted 2017-02-16; First posted 2017-04-21 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Septic Shock; Shock, Septic; Lactic Acidosis; Thiamine Deficiency
MeSH Terms: conditions — Shock, Septic; Acidosis, Lactic; Thiamine Deficiency | interventions — Thiamine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thiamine Supplementation Group (Experimental): Patients will receive 200mg thiamine in 50mL of 5% dextrose once daily for 7 days or until discharge from the intensive care unit.
  Interventions: Drug: Thiamine
- Placebo Group (Placebo Comparator): Patients will receive placebo (50mL 5% dextrose) once daily for 7 days or until discharge from the intensive care unit.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Thiamine
  Other Names: Vitamin B1
  Arms: Thiamine Supplementation Group
Drug: Placebos
  Other Names: 50mL 5% dextrose
  Arms: Placebo Group

SUMMARY:
To determine if intravenous thiamine would decrease the time to reversal of shock in patients with septic shock.

DETAILED DESCRIPTION:
Patients will be randomized to thiamine supplementation or placebo in a 1:1 ratio. Randomization will be done by the hospital pharmacy department whom will be the only unblinded participants. Patients will receive 200mg thiamine in 50mL of 5% dextrose or matching placebo (50mL 5% dextrose) once daily for 7 days or until discharge from the intensive care unit. The drug will be mixed by the pharmacy. Administration will be done in the patients room in the intensive care unit by the patient's assigned nurse. Blood will be collected on admission to the hospital in order to determine baseline lactate level and study eligibility. The measurement of lactate is standard of care in patients with sepsis. Thiamine level will be collected upon enrollment into the study. The ICU nurse or emergency room nurse taking care of the patient at the time of enrollment will draw the blood sample. Standard procedure for measuring thiamine levels will be maintained including protecting the blood sample from light and keeping it on ice while it is delivered to the lab. Serum lactate will be measured daily for 7 days or until discharge from the intensive care unit. The serial measurement of serum lactate is considered standard of care in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Sepsis (defined as presence of two or more SIRS criteria with documented or suspected infection)
* SIRS: Systemic Inflammatory Response Syndrome (SIRS) is the occurrence of at least two of the following criteria: temperature >38.0ºC or <36.0ºC, heart rate >90 beats/minute, respiratory rate >20 breaths/minute, white blood cell count >12,000 or <4000.
* Lactate >3mmol/L at the time of consent and randomization
* Hypotension (systolic blood pressure <90mmHg) after a >2L fluid bolus
* Vasopressor dependence (defined as the continuous infusion of norepinephrine, dopamine, phenylephrine, vasopressin or epinephrine.)

Exclusion Criteria:

* Known cirrhosis or chronic liver disease
* Current thiamine supplementation
* Clinical indication for thiamine (e.g. Alcohol abuse)
* Comfort measures only designation
* Inability to provide consent
* Other causes for lactate elevation (seizure, use of medications that can cause lactic acidosis such as metformin, linezolid and anti-retrovirals, carbon monoxide, known or suspected bowel or limb ischemia, cardiac arrest prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-05 (Actual); Primary Completion 2019-03-14 (Estimated); Study Completion 2019-03-14 (Estimated)

PRIMARY OUTCOMES:
Time to Reversal of Shock | 7 days
  Number of hours that the patient required vasopressors
Time to Normalization of Lactic Acidosis | 7 days

SECONDARY OUTCOMES:
ICU Mortality | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Death occurring during the ICU stay
ICU Length of Stay | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Number of days that the patient remains in the ICU after admission to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Jinesh Mehta, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No